CLINICAL TRIAL: NCT02604251
Title: A Prospective Randomized Clinical Study Evaluating the Safety and Efficacy of the KLOX BioPhotonic WoundGel System When Compared With Silicone Sheets in the Treatment of Surgical Wounds
Brief Title: Evaluation of the KLOX BioPhotonic WoundGel System in the Treatment of Surgical Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KLOX Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-K1002-P010
Record Dates: First submitted 2015-11-06; First posted 2015-11-13 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Surgical Wounds
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment with KLOX BioPhotonic WoundGel System (Experimental): One breast will be randomized to be treated with KLOX BioPhotonic WoundGel System.
  Interventions: Device: KLOX BioPhotonic WoundGel System
- Treatment with silicone sheets (Active Comparator): The second breast will be randomized to be treated with silicone sheets.
  Interventions: Device: Silicone sheets

INTERVENTIONS:
Device: KLOX BioPhotonic WoundGel System — Patients will then be re-randomized to one of the three comparisons: treatment starting on day 7 post-surgery, treatment starting on Day 21 post-surgery, or two consecutive treatments applied once weekly.
  Arms: Treatment with KLOX BioPhotonic WoundGel System
Device: Silicone sheets — Treatment of the surgical wounds with silicone sheets.
  Arms: Treatment with silicone sheets

SUMMARY:
This is a multicenter, randomized, prospective, controlled study in patients having bilateral breast reduction. Objectives of the study are to evaluate the safety and efficacy of the KLOX BioPhotonic WoundGel System compared with the ones of Silicone Sheets in the treatment of surgical wounds.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent form
2. Female patients, aged between 18 and 75 years old
3. Good general health, stable weight, free of systemic diseases such as diabetes, arthritis, HIV infection or genetic disorder that could influence the outcome of the treatment
4. Fitzpatrick skin type I to IV
5. Patients scheduled to go through bilateral breast reduction and expected to have newly formed post-surgery breast incisions of comparable length, located on comparable skin area
6. Patients able to understand, willing and able to comply with all study requirements
7. Patients must either be incapable of reproduction, or taking acceptable measures to prevent pregnancy and have a negative pregnancy test prior to participation in the Study
8. Females of childbearing potential must not be lactating at Study Screening and agree to use adequate contraceptive method during the Study

Exclusion Criteria:

1. Inability to understand the Study and its requirements or to give informed consent
2. Patient has participated in any other clinical study within 3 months prior to Study Screening and throughout the Study duration
3. Systemic antibiotic therapy or anti-inflammatory drugs or any other medication(s) that might interfere with healing within the last three months prior to Study Screening and throughout the Study duration
4. Current use of anticoagulants such as (but not limited to) warfarin, clopidogrel, enoxaparin or high doses of aspirin (> 162 mg daily)
5. Patient with current alcohol use or actively consuming drugs (addiction) as it may interfere with patient's ability to comply with Study procedures
6. Female patient pregnant, nursing or planning to become pregnant within the next 18 months
7. Patient is a current smoker or has been smoking or using nicotine product(s) in the last three months
8. Patient with known photosensitivity, taking drug(s) to treat photosensitivity, with concurrent disease (such as porphyria) or drug(s) (such as methotrexate or chloroquine) known to induce severe photosensitivity of the skin
9. Patients who are immunocompromised or taking immunosuppressive therapy
10. Any concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the Study investigational device
11. Patient has ongoing malignant disease of any type, active systemic, local skin infection or disease, autoimmune disease or any significant chronic disease which, in the opinion of the investigator, might interfere with the evaluation of the Study objectives or would result in non-compliance with the Study protocol
12. Patients with known hypersensitivity to pain medications
13. Patients with severe elastosis
14. Patients with severe or cystic acne on the area(s) to be treated
15. Presence of a metal stent or implant in the area(s) to be treated
16. Patients with derma resurfacing procedures or non-invasive skin-tightening procedures including medium/deep chemical peeling, microdermabrasion, laser therapy or prescription level glycolic acid treatment to the treatment area(s) within three months prior to Study Screening or during the Study
17. Patients anticipating the need for surgery or overnight hospitalization during the course of the Study
18. Patients with history of keloids or hypertrophic scars
19. Patients anticipating sun tanning bed or excessive sun exposure during the Study period
20. Patients with significant breast asymmetry that may result in asymmetrical operative incisions being made on the left and right breasts
21. Patients with breast asymmetry that may result in different post-operative tensions on the wounds of the left and right breasts
22. Patients having had surgery in the area to be incised within one year of Study Screening
23. Patients with tattoos in the areas of incisions
24. Patients with incisions that are actively bleeding
25. Patients with history of irradiated breast(s) in the area(s) to be treated.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Adverse Events, Serious Adverse Events and Device Incidents | 24 weeks
  Number of patients with adverse events, serious adverse events and device incidents

SECONDARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) | up to 24 weeks
  Assessment of the efficacy of the KLOX BioPhotonic WoundGel System and of Silicone Sheets by the patient and by the investigator via the POSAS
Vancouver Scar Scale (VSS) | up to 24 weeks
  Assessment of the efficacy of the KLOX BioPhotonic WoundGel System and of Silicone Sheets by the investigator via the VSS
Efficacy as assessed by blinded experts panel | up to 24 weeks
  Assessment of the efficacy of the KLOX BioPhotonic WoundGel System and of Silicone Sheets by a blinded experts committee
Ease of wound management | up to 24 weeks
  Patient's self-assessment of ease of wound management by a specific questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Victoria Park Medispa, Montreal, Quebec
  - Westmount Aesthetic Surgery Centre, Montreal, Quebec